CLINICAL TRIAL: NCT06005831
Title: Is Application of Uterine Fundus Pressure With a Sandbag Effective in Reduction of Cesarean Bleeding? A Prospective Case Control Stud
Brief Title: Uterine Fundus Pressure in Reduction of Cesarean Bleeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Firat University (Other)
Responsible Party: Principal Investigator, Mustafa YILMAZ, Firat University, Firat University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020/14-02
Record Dates: First submitted 2023-08-01; First posted 2023-08-23 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Postoperative Bleeding
Keywords: cesarean section; fundal pressure; postoperative bleeding; sandbag
MeSH Terms: conditions — Postoperative Hemorrhage

STUDY DESIGN:
Intervention Model Description: It is a prospective, randomized, controlled single-center study.
Masking Description: The 482 patients who had CS were divided into two groups, control group (n = 246), weighted group (n = 236) was randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sandbag (Other): Sandbag
  Interventions: Other: sandbag

INTERVENTIONS:
Other: sandbag — The standard sandbag used in our clinic, 20 × 20 × 3 cm3 in dimensions and 3 kg in weight

SUMMARY:
Uterine compression methods reduce the amount of postpartum bleeding. In our study, we investigated the effect of fundal pressure, which will be created by a sandbag placed on the abdomen, on reducing post-cesarean bleeding. Material and Methods: A total of 482 patients who delivered by cesarean section (CS) in the Obstetrics Clinic of Fırat University Faculty of Medicine between January 2021 and December 2021 were included in this prospective, randomized, single-center study.

DETAILED DESCRIPTION:
A total of 482 patients who gave birth by CS in the Obstetrics Clinic of Fırat University Faculty of Medicine between 1 January 2021 and 31 December 2021 were included in the study. Approval was obtained from the Ethics Committee of Fırat University for this prospective randomized single-center study (Ethics committee date = 15.10.2020; decision no = 2020/14-02). The 482 patients who had CS were divided into two groups, control group (n = 246), weighted group (n = 236) was randomized. Each patient was followed up in our obstetrics clinic until discharge from the hospital after surgery and the data were analyzed. The same techniques were used in all surgical procedures in order not to create differences in terms of surgical techniques and operation times that may affect intraoperative bleeding. However, to minimize inter-operator variations, surgical procedures were performed by operators with sufficient surgical experience.

The standard sandbag used in our clinic was 20 × 20 × 3 cm3 in dimensions and 3 kg in weight. Sandbags of the same standard were used for all patients. After the patient was taken to the patient's bed, the uterine fundus was palpated, and then the sandbag was placed on the abdomen, just above the fundus, in such a way as to apply pressure to the fundus. The sandbag was kept on the abdomen for approximately 6 hours. During this period, the patient was followed up frequently and care was taken not to change the position of the sandbag. Sandbags were removed just before our patients were mobilized (approximately 6 hours). The sandbag was placed on the same spot in each patient by the obstetric assistants in our author team. In addition, preoperative and postoperative follow-ups and data acquisition and storage were performed by the same team 2.1 Study Design

It is a prospective, randomized, controlled single-center study.

2.2 Inclusion Criteria

All cases with CS who had a live pregnancy after 24 weeks of gestation were included in the study.

2.3 Exclusion Criteria

* Invasion anomaly,
* Diagnosed with preeclampsia,
* Placenta previa cases,
* Hypertensive pregnant women receiving antihypertensive therapy,
* Diabetic pregnant women,
* Multiple pregnancies,
* Major hepatic, cardiac, renal, respiratory disorders
* Deep vein thrombosis during pregnancy,
* Receiving anticoagulant therapy
* Patients who developed atony and uterine rupture in the operating room,
* Suspected placental invasion
* Uterine balloon tamponade
* Arterial embolization
* Uterine and hypogastric artery ligation,
* Uterine compression sutures
* Intraoperative blood loss was estimated to be over 1000 mL during CS and who received intraoperative blood transfusion

2.4 Patient Selection

For randomization, patients were fully informed about the study while preparing for CS. Sandbags were placed in all cases included in the study after meeting the study criteria for between 1 January 2021 and 30 June 2021. Sandbags were not placed in the cases who met the study criteria and were included in the study between 1 July 2021 and 31 December 2021.2.5 Sampling Technique

Qualified participants who gave informed consent to participate in the study were randomly assigned to groups. Visual analog scale (VAS) was used for postoperative pain scoring at the 8th and 24th postoperative hours. The patient included in the study was randomized into control group or weighted group by another assistant doctor who did not participate in the CS and did not know about the patient.

2.6 Postoperative Monitoring

All cases were given 10 IU of oxytocin IV during CS, after prophylactic antibiotic therapy and placenta separation. After CS, 40 IU of oxytocin (Synpitan® forte ampule 5 IU, Deva, Istanbul, Turkey) was administered intravenously in 500 mL saline and at an infusion rate of 125 mL/hour. At the same time, 0.2-0.4 µg methylergonovine maleate (Methergine® ampule 0.2 µmg, Sandoz, Istanbul, Turkey) was given intravenously/intramuscularly in cases without hypertension. All patients were treated according to the postoperative protocol for CS performed in our obstetrics clinic. At the 8th and 24th hours postoperatively, the researchers determined the patient's hemoglobin (Hb) and hematocrit (Hct) concentrations and the amount of vaginal bleeding. In addition, the time of milk coming from the breast and VAS were performed. Patients with a postoperative Hb value of <7 g/dL received blood transfusion. Considering the risks of blood transfusion, blood transfusion is primarily planned in symptomatic patients with an Hct value of <20%, as stated in the bulletin of The American College of Obstetricians and Gynecologists (ACOG), but if the Hb is below 7 g/dL, it is hemodynamically stable and in asymptomatic patients, the treatment is individualized and alternative to transfusion, oral anti anemic or intravenous iron therapy is applied.

2.7 Determination of the Amount of Postoperative Blood Loss

Postoperative blood loss was determined by monitoring the pad and measuring the hemoglobin values at the 8th and 24th hours in all cases. Standard pads measuring 10 × 10 cm2 was used. The main advantage of this method of visually assessing blood loss is that it is a real-time assessment and allows the person accompanying the delivery to correlate it with the patient's clinical findings. However, significant differences between clinical evaluation and actual measurements have been clearly demonstrated in many studies has been reported that gravimetric blood loss estimation methods or serum lactate measurements can provide a more objective assessment of bleeding. It has been reported that visual and gravimetric blood loss estimation measurements show a high degree of bias and therefore their routine use cannot be recommended. On the other hand, it has been stated that colorimetric technology offers real-time measurement and has a high degree of correlation. For this reason, we used the preoperatively and postoperatively at the 8th and 24th hours hemoglobin values. Postpartum anemia was defined as hemoglobin concentration (Hb) <10 g/dL in the postpartum period.

ELIGIBILITY:
Inclusion Criteria

All cases with CS who had a live pregnancy after 24 weeks of gestation were included in the study.

Exclusion Criteria

* Invasion anomaly,
* Diagnosed with preeclampsia,
* Placenta previa cases,
* Hypertensive pregnant women receiving antihypertensive therapy,
* Diabetic pregnant women,
* Multiple pregnancies,
* Major hepatic, cardiac, renal, respiratory disorders
* Deep vein thrombosis during pregnancy,
* Receiving anticoagulant therapy
* Patients who developed atony and uterine rupture in the operating room,
* Suspected placental invasion
* Uterine balloon tamponade
* Arterial embolization
* Uterine and hypogastric artery ligation,
* Uterine compression sutures
* Intraoperative blood loss was estimated to be over 1000 mL during CS and who received intraoperative blood transfusion

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Uterine compression methods reduce the amount of postpartum bleeding
Enrollment: 482 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Whether the fundal pressure created by the sandbag placed on the abdomen has an effect on reducing post-cesarean bleeding. | 24 hours
  Whether the fundal pressure created by the sandbag placed on the abdomen has an effect on reducing post-cesarean bleeding.

CONTACTS AND LOCATIONS:
Overall Officials: Sehmus Pala, Study Chair — University of Firat
Locations (1):
- Firat University Faculty of Medicine, Elâzığ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No